CLINICAL TRIAL: NCT03506269
Title: Perception and Knowledge About Menopause Among Pakistani Woman
Status: Completed | Type: Observational
Sponsor: OBS Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS-Tibol-001
Record Dates: First submitted 2018-04-11; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted to find out perception and knowledge about Menopause among Pakistani Woman.

DETAILED DESCRIPTION:
The survey for was conducted in various location and clinics all over Pakistan. 1200 numbers of questionnaires were distributed of which 910 numbers responded from 1st January 2018 to 28th February 2018. Those who agreed to be part of study where ask a self-structured questionnaire related to awareness and symptoms of menopause. Data was analyzed using SPSS Version 23.0. Frequencies were calculated for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 35 to 55
* Oral Informed consent

Exclusion Criteria:

* None

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Females aged 35 to 55 were enrolled after taking their oral informed consent. The survey for was conducted in various location and clinics all over Pakistan. 1200 numbers of questionnaires were distributed of which 910 numbers responded from 1st January 2018 to 28th February 2018. Those who agreed to be part of study where ask a self-structured questionnaire related to awareness and symptoms of menopause.
Sampling Method: Non-Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
To Find Perception and Knowledge of Menopause in Pakistani Woman | 0-28 days
  To find perception and knowledge of Menopause in Pakistani woman based on self-structured questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Faizan Shaukat, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No